CLINICAL TRIAL: NCT03980912
Title: Clinical Diagnostic Validation of the LiverFASt Test and the Associated Fibrosis Staging Scores for Activity/Inflammation and Steatosis as Compared to Liver Tissue Pathology Via Liver Biopsy
Brief Title: Validation of the LiverFASt Test and the Associated Fibrosis Staging Scores Compared to Liver Tissue Pathology Via Liver Biopsy
Status: Withdrawn | Type: Observational
Why Stopped: created a new protocol with a new study design
Sponsor: Fibronostics USA, Inc (Other)
Collaborators: OBVIO HEALTH USA, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: OBVIO-FIB-001
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: NAFLD; NASH
Keywords: LiverFASt; Fibrosis; Steatosis; Activity; Liver Biopsy; Algorithm; LiverFASt select; Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Fatty Liver; Motor Activity; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: LiverFASt — LiverFASt™ is a blood based diagnostic test utilizing a patented algorithm to determine presence and the progression of liver disease. The test is non-invasive, simple, and less expensive than liver biopsy or liver imaging.

SUMMARY:
This study is to assess the diagnostic performance of the LiverFASt Test for assessing fibrosis staging scores compared to the assessment of liver tissue pathology from liver biopsy.

DETAILED DESCRIPTION:
Chronic liver diseases (CLDs), such as chronic viral hepatitis, nonalcoholic fatty liver diseases (NAFLD) and nonalcoholic steatohepatitis (NASH), are a leading cause of morbidity and mortality globally and usually develops over many years. The prevalence of NAFLD has increased in recent years (15% in 2005 to 25% in 2010). As, approximately 20% of NAFLD cases develop NASH, the associated increase in NASH during the same period is to be expected (33% in 2005 to 59.1% in 2010).

The risk of liver-related mortality increases exponentially with increase in fibrosis stage. As the progression from NAFLD to NASH is associated with progressive liver fibrosis, the prognosis for NASH is worse than it is for NAFLD, and results in an increased risk of cirrhosis, hepatocellular carcinoma (HCC) and death from liver related causes. As a result, staging of liver fibrosis is essential in determining the prognosis and optimal treatment for patients with NASH. Furthermore, evaluation of fibrosis in NAFLD patients can help refine treatment options designed to prevent the progression to NASH. Currently, liver biopsy is the gold standard for staging liver fibrosis. However, liver biopsy is invasive, expensive and prone to sampling error. Developing, safe and easily accessible noninvasive modalities to accurately evaluate fibrosis stage of NAFLD and NASH is of utmost importance in clinical practice. The use of non-invasive biomarkers of liver fibrosis are needed in the general population setting.

LiverFASt is a non-invasive diagnostic and staging tool, which has been developed as an alternative to liver biopsy. It is a reliable, and reproducible tool which provides grading or staging of the three elementary features of NASH: steatosis, inflammatory activity and fibrosis. The main aim of this study is to evaluate the diagnostic value of LiverFASt as a non-invasive biopsy-proven assessment of fatty liver disease.

Early liver disease detection allows patients treatment options for a healthier and productive life. Once liver disease progresses to cirrhosis or cancer, treatment options are limited and expensive. Reducing the almost $2Billion dollar liver disease economic burden to the United States, requires a breakthrough technology, which brings diagnosis to the patient.

Current liver disease diagnosis devices are dependent on fixed facilities, which utilize ultrasound, CT scan, MRI or biopsy sampling with pathology analysis. The dependency on fixed facility diagnostic procedures introduces barriers to patients receiving early detection. While it is known that early detection, wellness and cost effectiveness mitigate these realities, and many trends today in diagnostics are pushing greater early access to the patients, providers limit screening and detection to patients for which the procedure meets the cost-benefit in the ever-evolving value-based healthcare system. Additionally, requiring patients to travel to radiology or laboratory facilities introduces adherence issues.

Fibronostics breaks through the burden to serve patients. By empowering their providers with diagnostic tools within the clinic, the ability to ensure screening and diagnostic adherence is eliminated, and the ease for early detection profoundly shifts the $2B economic burden. For example, the Veterans Health Affairs estimates that 50,000 veterans a year are undiagnosed for Hep C.

Fibronostics diagnostic tool fits into a backpack, which allows a broader reach to underserved patients, and supports the Veterans Health Affairs Mobile Health Provider Program, which is designed to equip VA health care providers with technologies to deliver health care to Veterans homes. To date there is no liver diagnostic device which can serve the broad United States population and shift the growing economic burden.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years old, inclusive
* Male or Female
* Liver patients who are scheduled to undergo, or have recently undergone, a medically indicated liver biopsy. Patients with a prior biopsy may be included under the following conditions:

  * The biopsy was performed within the 3 months prior to enrollment
  * A full report is available, including degree of Fibrosis, Activity and Steatosis or residual liver tissue is available for additional review.
* Have a full component of biomarkers available for analysis from a blood sample obtained within 3 months of the date of the biopsy. Participants without a full component of biomarkers may be included if an additional sample for analysis of the missing biomarkers can be obtained within 3 months of the date of the biopsy.

  * Required biomarkers include: α2-macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin, y-glutamyl transpeptidase (GGT), alanine aminotransferase (ALT), aspartate transaminase (AST), triglycerides, cholesterol, and fasting glucose, collected within 3 months
* Willing and able to allow access to requested data and who were informed and signed the consent form

Exclusion Criteria:

* Known psychiatric conditions
* Patients who may be uncooperative with the sample collection procedures
* Severe coagulopathy or infection of the hepatic bed
* Extrahepatic biliary obstruction
* Severe cardiovascular disease and/or renal failure
* Malignancy, except for resolved basal-cell carcinoma
* Previous liver transplant
* Suffering with a terminal illness or any other conditions or diseases that the investigator considers inappropriate for study participation

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include approximately 200 men and women residing in the United States, who are between the ages of 18-80 years. Participants will be liver patients who have undergone liver biopsy within the three months prior to enrollment or are scheduled to undergo a medically indicated liver biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of the LiverFASt test for NAFLD | Baseline
  Diagnostic performance of the LiverFASt Test for NAFLD resulting from liver biopsy based on percent diagnostic agreement using the thresholds of clinical significance outlined below.
Diagnostic Performance of the LiverFASt test for NAFLD | Baseline
  Diagnostic performance of the LiverFASt Test for NAFLD resulting from liver biopsy based on percent diagnostic specificity using the thresholds of clinical significance outlined below.
Diagnostic Performance of the LiverFASt test for NAFLD | Baseline
  Diagnostic performance of the LiverFASt Test for NAFLD resulting from liver biopsy based on percent diagnostic sensitivity using the thresholds of clinical significance outlined below.
Diagnostic Performance of the LiverFASt test for NAFLD | Baseline
  Diagnostic performance of the LiverFASt Test for NAFLD resulting from liver biopsy based on percent diagnostic accuracy using the thresholds of clinical significance outlined below.

SECONDARY OUTCOMES:
Diagnostic Performance of the LiverFASt test for NASH | Baseline
  Diagnostic Performance of LiverFASt Test in NASH compared to histopathology
Diagnostic Performance of the LiverFASt test for NASH | Baseline
  Performance of the test in determining the degree of Fibrosis, Activity and Steatosis compared to histopathology resulting from liver biopsy using percent composite score agreement
Diagnostic Performance of the LiverFASt test for NASH | Baseline
  Performance of the test in determining the degree of Fibrosis, Activity and Steatosis compared to histopathology resulting from liver biopsy using diagnostic stage-specific percent agreement.
Diagnostic Performance of the LiverFASt test for NASH | Baseline
  Performance of the test in determining the degree of Fibrosis, Activity and Steatosis compared to histopathology resulting from liver biopsy using deviation in individual composite score
Diagnostic Performance of the LiverFASt test for NASH | Baseline
  Performance of the test in determining the degree of Fibrosis, Activity and Steatosis compared to histopathology resulting from liver biopsy using sensitivity, specificity and accuracy for a stage score basis

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — OBVIO HEALTH USA, Inc.
Locations (1):
- ObvioHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Fibronostics — https://www.fibronostics.com/